CLINICAL TRIAL: NCT06912425
Title: Effects of an Exercise Program and a Protein Controlled Diet Using an Educational Intervention on Biochemical Parameters, Muscle Strength and Body Composition in Patients With Stage G1 and G2 CKD
Brief Title: Effects of an Exercise and Diet Program on Biochemistry and Body Composition in Patients With CKD in G1 and G2 Stages
Acronym: Renactivity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Ana Patricia Zepeda Salvador, Effects of an Exercise and Diet Program on Biochemistry and Body Composition in Patients With CKD in G1 and G2 Stages, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 97/HRCG-JAL/2023; AGAF2024/2 (Other: Universidad de Guadalajara)
Record Dates: First submitted 2024-06-17; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Kidney Diseases; Diet, Healthy; Dietary Habits; Exercise; Kidney Disease; Educational; Body Composition; Renal Failure , Chronic
Keywords: health belief model; kidney chronic disease; exercise; diet
MeSH Terms: conditions — Kidney Diseases; Feeding Behavior; Motor Activity; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Humans with CKD in stages 1 and 2
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supervised Exercise Intervention Group (Experimental): This group will be assigned a personalized exercise program designed by the researchers, specialists in kidney disease training. Participants will be assigned to the supervised exercise intervention through a randomization process, ensuring a homogeneous sample
  Interventions: Behavioral: Health prevention.
- Exercise Based on KDIGO Recommendations (Experimental): To this group will be assigned KDIGO exercise.
  This group will be assigned exercise based on KDIGO recommendations. They will be provided with an exercise template according to KDIGO guidelines, without further exercise planning. Additionally, they will receive a protein-controlled diet along with an educational intervention.
  Interventions: Behavioral: Health prevention.

INTERVENTIONS:
Behavioral: Health prevention. — Unlike other projects, this study focuses on an underexplored area in exercise and kidney disease research. Typically, exercise recommendations are directed toward individuals undergoing hemodialysis or peritoneal dialysis. However, in the early stages of the disease, when the kidneys begin to show alterations, there is no established safe training protocol as a preventive measure. This clinical trial will fill that gap by providing references for an exercise program specifically designed for individuals in the early stages of kidney disease. The main objective will be to compare two different exercise strategies to determine potential benefits for renal health.

SUMMARY:
How Exercise, a Controlled Diet and Education Improve the Health of People with Early-Stage Renal Failure: A Study at Ciudad Guzmán Hospital

DETAILED DESCRIPTION:
Chronic kidney disease has a high mortality rate per year, which has led to the search for different intervention strategies to improve adherence to treatment and the promotion of healthy behaviors such as diet and exercise. The latter has been little explored in early stages (G1 and G2) even though its implementation can have an impact on the biochemical parameters of patients and delay their progression. Exercise represents a non-pharmacological, non-invasive, and cost-effective method in health promotion, as it can reduce biomarkers of inflammation such as C-reactive protein, interleukin-6, tumor necrosis factor-α, among others. Despite this, statistics show that 27% of adults in the world do not do the 150 minutes of exercise per week recommended by the World Health Organization (WHO). Regarding medical indications for exercise, there is a prevailing resistance in the medical community regarding its recommendation, given that proteinuria and/or changes in blood pressure linked to this activity are considered to have an impact on renal function. Existing exercise recommendations and proposals are focused on patients on peritoneal dialysis or hemodialysis. One of the most widespread in this patient population are the recommendations made by the WHO for older people with chronic conditions, and more specifically, there are the kidney disease: Improving Global Outcomes (KDIGO) guidelines, however, both give general recommendations, and it has been pointed out as a point of opportunity to explore exercise in this population. The published interventions are limited and do not include biochemical parameters in most of them, nor the physical aptitudes of the patients when performing exercise. On the other hand, it has been identified that the reduction of complications in these patients is associated with healthy behaviors, such as exercise, greater adherence to diet and pharmacological treatment. Several structural barriers have been detected, such as ideological barriers, beliefs, access to treatments, among others, which influence patients' lack of adherence to the plans. Considering the above, the aim of the present research will be to analyze the effects of an exercise program and a protein-controlled diet using an educational intervention on biochemical parameters, muscle strength and body composition in patients with chronic kidney disease in stage G1 and G2. The intervention will be for 3 months and will have two groups: one will follow an exercise program designed for each participant; the second group will follow the exercise recommendation proposed by the KDIGO 2022 guidelines. Both groups will have a personalized dietary plan, educational sessions, body composition and muscle strength assessment monthly. Biochemical parameters such as: creatinine, cystatin C, glucose, urea, urinary sediment, among others, will be evaluated at the beginning and at the end of the intervention to compare changes. Regarding adherence to both the exercise program and the diet, we will seek to reduce the patients' structural barriers by means of educational sessions based on the health belief model (HBM). Topics such as: knowledge of the disease, culinary techniques, barriers that prevent adherence to treatment, among others, will be taught. This project is expected to generate novel knowledge regarding the impact of an educational intervention combined with exercise in patients with chronic kidney disease in early stages. This information may be relevant to guide recommendations in clinical practice guidelines, in addition to promoting the adoption of healthy behaviors such as structured exercise.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of CKD by the physician in G1 and G2
* Who meet the requirements of normal or decreased filtration rate according to:
* G1: ≥ 90 or G2: 60-89 mL/ min/ 1.73m2
* Alterations in the urinary sediment (cellular cylinders of any type, dysmorphic erythrocytes).
* Confirmation of damage by renal ultrasound (Decreased renal size, thinning of the renal cortex, increased echogenicity of the parenchyma, poor differentiation between the renal cortex and sinus, renal cysts suggestive of cortical or medullary changes).
* Men and women between 18 and 65 years old
* Control of baseline pathologies (glycosylated hemoglobin less than 9%, blood pressure no higher than 140/90mmHg).
* Patients who agree to participate in the study and sign the informed consent form.
* Patients who have no limitations to perform the exercises.
* If participants have diagnosed diabetes or hypertension, who are on medication and under regular internal medicine or nephrology treatment.
* Male and female patients, including those who are illiterate but can be accompanied in the initial sessions to sign the informed consent form.
* All participants, even those who do not have a mobile device, will be provided with an exercise and nutrition guide so that they do not have any limitations when carrying out the activities.

Exclusion Criteria:

* Stages 3, 4 and 5
* Children under 18 years of age
* Patients who, due to their place of origin, find it difficult to travel to the sessions.
* Diabetes Mellitus in uncontrolled (Glycated Hemoglobin >9 %)
* Those who have lost their sight
* Presence of uremic alterations such as uremic encephalopathy.
* Who present unstable blood pressure with blood pressure levels above 140/90mmHg, patients showing sustained blood pressure elevations above 140/90 will be discontinued from the study.
* Peripheral vascular disease of all types (Peripheral Arterial Disease (PAD), Deep Vein Thrombosis (DVT), Chronic Venous Disease (CVD), Abdominal Aortic Aneurysm (AAA), Buerger's Phenomenon (Thromboangiitis Obliterans), Kawasaki Disease).
* Failure to sign the informed consent form

Elimination Criteria:

* Injury, discomfort that makes reincorporation impossible.
* Patients who have decided to abandon the study
* Patients who do not attend 2 of the face-to-face sessions, those who do not attend two of their sessions will be taken into consideration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-10-28 (Estimated)

PRIMARY OUTCOMES:
Changes in total cholesterol | changes from baseline to week 12
  Total cholesterol: A decrease in values is expected, taking as reference a normal range of <200 mg/dL. This will indicate a better outcome of the intervention. A change obtained from week 1 to week 12 is expected.
Changes in HDL cholesterol | Changes from baseline measurement to week 12
  HDL cholesterol: An increase in its values is expected, with a normal range of >40 mg/dL. The increase will mean better cardiovascular outcomes. Change is expected from week 1 to week 12.
LDL cholesterol changes | Changes from basal levels up to week 12
  LDL cholesterol: A reduction in its levels is expected, considering a reference value <100 mg/dL. The decrease will mean better cardiovascular outcomes. Evaluation from week 1 to week 12.
Changes in triglycerides levels | Changes from baseline measurement to week 12
  Triglycerides: a decrease in values is expected, with a reference range <150 mg/dL. The decrease will mean better cardiovascular outcomes
Changes in albumin level | Changes from baseline levels to week 12
  Albumin: An increase in its values is anticipated, with a normal range of 3.5-5 g/dL. Its increase will be considered an adequate nutritional parameter and a decrease of inflammatory marker. Evaluation from week 1 to week 12.
Changes in vitamin D levels | Changes from baseline levels at week 12
  Vitamina D (25-hidroxivitamina D o 25(OH)D): Se espera un aumento de los valores, tomando como referencia un rango de 30-50 ng/mL. Evaluación de la semana 1 a la semana 12.
Changes in insulin levels | Changes from baseline to week 12
  Insulin: Changes in its values will be analyzed, considering a reference range of 2-25 U/mL. Its increase will be considered a favorable result. Evaluation from week 1 to week 12.
Changes in Creatina fosfoquinasa (CK total) | Changes from baseline to week 12
  Creatine Phosphokinase (Total CK): Values are expected to be maintained or increased as a result of adaptation to exercise, with a reference range of 26-192 U/L. Evaluation from week 1 to week 12.
Changes in the quality of life questionnaire KDQOL-SF | Changes in initial (week 1) and final responses (week 12)
  Kidney Disease Quality of Life: Improvements are expected in the questionnaire score, ranging from 0 (lowest quality of life) to 100 (highest quality of life). Assessment from week 1 to week 12.
Changes in the answers to the questionnaire "Knowledge of the disease". | changes in initial (week 1) and final responses (week 12)
  Questionnaire "Knowledge of the disease": The changes in the correct answers to the 13 items will be analyzed by means of a score based on the Likert scale. Evaluation from week 1 to week 12.
Changes in the answers to the questionnaire - Opinion on the disease | changes in initial (week 1) and final responses (week 12)
  Opinión sobre la enfermedad: Se evaluarán los cambios en la percepción de los participantes sobre su enfermedad, determinando su grado de acuerdo o desacuerdo con diferentes afirmaciones.
Adherence in exercise frequency | initial changes (week 1) and final changes (week 12)
  Exercise frequency: It will be measured by self-reporting, recording the number of weekly sessions and the duration of each one. A greater number of sessions will be considered a better indicator of results. Evaluation from week 1 to week 12.
Changes in grip strength | changes from the baseline measurement (week 1) to the final week (week 12)
  Grasping grip strength (dynamometer): An increase in dominant hand grip strength, expressed in kilograms, is expected. Ideal values are >25 kg, but in this population improvement over baseline measurement will be considered. Assessment from week 1 to week 12.

SECONDARY OUTCOMES:
Changes in fat mass | Comparative changes from baseline (week 1) to final measurement (week 12)
  Reduction of fat mass: It will be evaluated by electrical bioimpedance (InBody®), comparing the baseline measurement with the final measurement at week 12. A healthy body fat percentage will be taken as a reference point: ≤25% in women and ≤15% in men.
Muscle mass changes | Comparative changes from baseline (week 1) to final measurement (week 12)
  Increase in muscle mass: It will be analyzed through electrical bioimpedance (InBody®), considering an increase in relation to healthy reference values: ≥35% in men and ≥25% in women. Initial and final values (week 12) will be compared.
Changes in body mass index | Comparative changes from baseline (week 1) to final measurement (week 12)
  Body Mass Index (BMI): BMI changes in overweight patients will be evaluated, taking a healthy range of 20-25 kg/m² as a reference.
Changes in the responses to the questionnaire "frequency of food consumption for the Mexican population" | changes in responses to the questionnaire "food consumption frequency for the mexican population" comparing initial (week 1) and final (week 12) responses
  Increase in fruit and vegetable foods and decrease in processed foods, evaluated with the food consumption frequency questionnaire for the Mexican population.
Changes in visceral fat | Changes from baseline measurement (week 1) to final measurement (week 12)
  Changes in visceral fat measured from week 1 to week 12 by InBody bioimpedance scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Universitario del Sur, Ciudad Guzmán, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Body composition, biochemical parameters, muscle strength and food consumption frequency results.

REFERENCES:
- [Background] Ash S, Campbell KL, Bogard J, Millichamp A. Nutrition prescription to achieve positive outcomes in chronic kidney disease: a systematic review. Nutrients. 2014 Jan 22;6(1):416-51. doi: 10.3390/nu6010416. PMID 24451311